CLINICAL TRIAL: NCT05736926
Title: Anal Fissure Among Survivors of COVID-19 Virus Infection, Risk Factors and Outcome. A Single Center Experience.
Brief Title: Anal Fissure Among Survivors of COVID-19 Virus Infection.
Status: Completed | Type: Observational
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ahmad Sakr, consultant and lecturer of general surgery, Mansoura University
Other Study IDs: 1234
Record Dates: First submitted 2023-02-18; First posted 2023-02-21 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Anal Fissure; Corona Virus Infection
MeSH Terms: conditions — Fissure in Ano; Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background Anal fissure is one of the most common anorectal problems. After an outbreak of coronavirus disease (COVID-19) has rapidly spread from China to almost all over the world, it nearly affected all countries. In spite of its typical presentation in the form of fever, cough, myalgia, fatigue and pneumonia, other GIT manifestations were reported. We found some of COVID-19 survivors who had complained from anal fissure problem. The aim of this study was to report the prevalence of acute anal fissure among COVID-19 patients, its possible risk factors and outcome.

Methods This is a retrospective cross-sectional study which was conducted over three months from the start of September 2020 to the end of November 2020 at Mansoura university isolation hospital, on COVID-19 patients' who were diagnosed with anal fissure. Those who survived and were discharged home safely were telephone called to pick up whether they suffered from any symptoms of anal pain, difficulty in defecation suggesting anal fissure, in order to identify their outcomes, the risk factors for anal fissure development and how they were managed.

Results A total of 176 patients were enrolled in this study. Patients were categorized into two groups. The first group included patients who developed anal fissure (n=65) and the 2nd group included patients who did not develop anal fissure (n=111). No significant difference was noted in demographic data apart from the age which was younger in the fissure group. The incidence of anal fissure was 36.9% of total population. The majority of patients' anal fissure problem resolved spontaneously after patients improved from the COVID symptoms without receiving any treatment (43.1%).

Conclusion Anal fissure is quite common problem after COVID-19. Young and middle age patients are more vulnerable to develop anal fissure after COVID-19 infection.

DETAILED DESCRIPTION:
Methods Study design This is a retrospective cross-sectional study which was conducted over three months from the start of September 2020 to the end of November 2020 at Mansoura university isolation hospital, on COVID-19 patients' who were diagnosed to have anal fissure. Mansoura isolation hospital is a tertiary referral center that admits COVID -19 patients. Patient who had experienced any symptoms that suggests COVID-19 infection and their nasal swab tested PCR positive were admitted. Also patients with CT chest findings that suggest COVID-19 infection were admitted.

The study protocol was approved by the Institutional Review Board (IRB) of Mansoura University (IRB No. R.21.07.1383). Informed consents were obtained from the patients.

Eligibility criteria Patients of both genders aging between 20-70 years with or without associated co-morbidities who received treatment for COVID-19 infection, were discharged home safely, and presented with anal fissure during the follow up were included. Patients who didn't experience anal pain or anal fissure, and patients who died were excluded from this study.

Patient interview By checking the Electronic medical records (EMR) during those 3 months, all patients' data was addressed and those who survived and were discharged home safely were telephone called to pick up whether they suffered from any symptoms of anal pain, difficulty in defecation suggesting anal fissure. Trying to identify their outcomes, the risk factors for anal fissure development and how they were managed. We telephoned about 350 patients, 176 replied to us while 174 didn't answer.

Those who suffered from anal pain problems were advised to come to our colorectal outpatient clinic (OPC) to be examined to make sure of the diagnosis. But, because of the pandemic situation, no patient came to the OPC. Further telephone calls were conducted to those who were diagnosed with anal fissure to ask about their outcomes, to pick up how many of them were managed medically or their symptoms resolved spontaneously or needed surgical interference.

All patient recorded data including; age, sex, the associated co-morbidities, and the degree of severity of infection, respiratory or GIT symptoms and the need for oxygen therapy were collected. Other symptoms as fever, loss of smell and/or taste sensation, constipation or diarrhea and also the duration of these symptoms were checked. Additionally, the investigations that were conducted either laboratory or radiological.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders
* Aging between 20-70 years
* With or without associated co-morbidities
* Those who received treatment for COVID-19 infection, were discharged home safely, Those who presented with anal fissure during the follow up were included.

Exclusion Criteria:

* Patients who didn't experience anal pain or anal fissure,
* Patients who died were excluded from this study.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All COVID-19 survivors who developed anal fissure
Sampling Method: Probability Sample
Enrollment: 176 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
incidence of anal fissure among covid -19 survivors | 6 months
  how many patients developed anal fissure among total patients

SECONDARY OUTCOMES:
risk factors associated with development of anal fissure | 6 months - 1year
  possible causes of fissure among this group

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmad, Al Mansurah, Egypt